CLINICAL TRIAL: NCT02385760
Title: A Multi-centre, Double-blind, Randomized, Parallel Group, Placebo Controlled Efficacy and Safety Study of Oral CTX-4430 for the Treatment of Moderate to Severe Facial Acne Vulgaris
Brief Title: CTX-4430 for the Treatment of Moderate to Severe Facial Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celtaxsys, Inc. (Other)
Collaborators: Clinical Network Services (CNS) Pty Ltd (Industry); Celtaxsys Aus Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTX-4430-AV-201
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Acne Vulgaris
Keywords: Facial Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — acebilustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): CTX-4430 oral capsule, 100 mg, once-daily for 12 weeks
  Interventions: Drug: CTX-4430
- Placebo (Placebo Comparator): Placebo: identical oral capsule, without active ingredient, once-daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CTX-4430
  Arms: Active
Drug: Placebo
  Arms: Placebo

SUMMARY:
A multi-centre, double-blind, randomized, parallel group, placebo controlled efficacy and safety study of oral CTX-4430 for the treatment of moderate to severe facial acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

1. Must provide Informed consent.
2. Male or female aged 16 to 44 inclusive.
3. Moderate to severe facial acne vulgaris as defined in the protocol.

Exclusion Criteria:

1. Positive testing for HIV, HBsAg, or hepatitis C virus (HCV).
2. Females who are pregnant, lactating, or planning to become pregnant during the study.
3. Any systemic medical condition which, in the opinion of the investigator, would put the participant at risk by participation in the study.
4. Any systemic or dermatologic disorder that, in the opinion of the investigator will interfere with the assessment of the study endpoints (e.g. psoriasis).
5. Concurrent or previous use of an investigational drug or device within 30 days prior to screening.
6. The presence of acne conglobata, acne fulminans, secondary acne, or nodulocystic acne.
7. The presence of known or suspicious unresolved dermatological cancerous or pre-cancerous lesions.
8. Hypersensitivity or idiosyncratic reaction to compounds related to CTX-4430 or any of its components.

Ages: 16 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Efficacy as measured by inflammatory lesion counts | 12 weeks
  Change from baseline in inflammatory lesion count after 12 weeks of treatment as compared to placebo.
Safety as measured by the incidence of treatment emergent adverse events | 12 weeks
  Incidence of treatment emergent adverse events as compared to placebo.

SECONDARY OUTCOMES:
Efficacy as measured by Investigator Global Assessment (IGA) | 12 weeks
  The proportion of participants achieving Grade 0 or 1 with a two grade improvement in the IGA from baseline to the end of the 12 weeks of treatment as compared to placebo.
Efficacy as measured by non-inflammatory lesion counts | 12 weeks
  Change from baseline in non-inflammatory lesion counts after 12 weeks of treatment as compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda J Spelman, MB BS, FACD, Principal Investigator — Veracity Clinical Research
Locations (10):
- Australia (8):
  - Clinical Trials Woden Dermatology, Phillip, Australian Capital Territory
  - St George Dermatology, Kogarah, New South Wales
  - Central Sydney Dermatology, Sydney, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Siller Medical, Brisbane, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - Skin and Cancer Foundation, Carlton, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- New Zealand (2):
  - Optimal Clinical Trials, Auckland
  - Clinical Trials New Zealand, Hamilton